CLINICAL TRIAL: NCT04844684
Title: Link Between the Metabolism of Cortisol and Bile Acids in Obese Patients Before and After Bariatric Surgery
Brief Title: Evaluation of Cortisol and Bile Acids Metabolism in Obese Patients
Acronym: CORTABO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_77; 2020-A03176-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: Cortisol; Bile acids; Obesity; Bariatric surgery; Insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood (EDTA 3 mL), serum, 24 hours urine (before RYGB, 1 month and 1 year after RYGB, liver tissue, adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese/non-diabetic patients undergoing gastric bypass surgery
  Interventions: Other: Blood and urine collection

INTERVENTIONS:
Other: Blood and urine collection — Blood sampling urine collections before RYGP and 1 month and 1 year after.

SUMMARY:
Bariatric surgery is currently the most efficient treatment for obesity. The sustained weight loss and metabolic improvement seen following Roux-en-Y gastric bypass (RYGB), is explained partly by modifications in hormones including bile acids (BA). After RYGB, an increased total BA pool and a reduction in hepatic cortisol exposure is observed. Hydroxysteroid 11-β dehydrogenase 1 (HSD11B1), steroid 5α-reductases (SRD5A), and steroid 5β-reductases, AKR1D1 (also a BA metabolizing enzyme), are three enzymes involved in the metabolism of cortisol in the liver and are known to participate in metabolic syndrome. Their activity has been shown to be decreased after RYGB. Interestingly, the mechanisms explaining the modification of hepatic cortisol exposure and the activity of theses enzymes after RYGB are unknown. In view of the few data suggesting a link between cortisol metabolism and bile acids, this work aim to study and characterize this link in a context of RYBP

ELIGIBILITY:
Inclusion Criteria:

* Non-menopausal women
* BMI between 35 and 50 kg/m² included
* Social insured
* Ability to give consent

Exclusion Criteria:

* moderate and severe kidney insufficiency
* hepatic insufficiency
* known gallbladder lithiasis
* history of cholecystectomy or cholecystectomy planned during the gastric bypass
* history of bariatric surgery except gastric band and gastric balloon
* history of type 1
* treatment interfering with the cortisol metabolism: taking oral or inhaled glucocorticoids within the last 6 months
* treatment by BA as ursodeoxycholic acid, bile acids sequester, statin, fibrate stopped less than 4 weeks ago

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women obese patient
Study Population: Patients admitted for bariatric surgery in the department of endocrine surgery at Lille University Hospital
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between the variations of urinary cortisol metabolites and plasmatic total BA level before and after RYGB | At 1 year

SECONDARY OUTCOMES:
Urinary cortisol metabolite profile modification | At 1 month after RYGP, at 1 year after RYGP
Urinary and plasmatic BA profile modification | At 1 month after RYGP, at 1 year after RYGP
Correlation between the variations of cortisol metabolites and the variations of metabolic parameters 1 year after gastric bypass | at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie ESPIARD, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Huriez - Service d'endocrinologie, diabétologie, nutrition et métabolisme, Lille, France